CLINICAL TRIAL: NCT02223065
Title: A Bioequivalence Study of Fixed-dose Combination Tablet of 5 Milligrams Saxagliptin/10 Milligrams Dapagliflozin Relative to Their Respective Individual Components Coadministered to Healthy Subjects in the Fasted State
Brief Title: Bioequivalence Study Coadministered to Healthy Subjects in the Fasted State
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CV181-364
Record Dates: First submitted 2014-08-19; First posted 2014-08-22 (Estimated); Results first posted 2016-04-27 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-03

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — saxagliptin; dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment A (Experimental): Single oral dose of saxagliptin tablet coadministered with dapagliflozin tablet
  Interventions: Drug: Saxagliptin; Drug: Dapagliflozin
- Treatment B (Experimental): Single oral dose of FDC (fixed-dose combination) tablet
  Interventions: Drug: Saxagliptin; Drug: Dapagliflozin

INTERVENTIONS:
Drug: Saxagliptin
  Other Names: Onglyza
Drug: Dapagliflozin
  Other Names: Farxiga in the United States; Forxiga in other countries

SUMMARY:
The purpose of this study is to demonstrate bioequivalence of coadministered drugs on healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form

   * Signed written informed consent must be obtained from the subjects in accordance with requirements of the study center's IRB or IEC before the initiation of any protocol-required procedures.
2. Target Population

   * Healthy subjects as determined by no clinically significant deviation from normal in medical history, psychiatric history, physical examination findings, vital sign measurements, 12-lead ECG measurements, physical measurements, and clinical laboratory test results.
3. Age and Reproductive Status

   * Males and females, ages 19 to 55 years, inclusive. To extent possible, the distribution of men and women between the sequences will be balanced
   * Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of study drug.
   * Women must not be breastfeeding. d) WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drugs saxagliptin and dapagliflozin plus 5 half lives of study drug dapagliflozin (the longer half life between the 2 drugs; 3 days) for a total of 3 days following treatment completion.

     e) Men who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drugs saxagliptin and dapagliflozin plus 5 half lives of dapagliflozin (the longer half life between the 2 drugs; 3 days) for a total of 3 days following treatment completion.

     f) Azoospermic males and WOCBP who are continuously not heterosexually active are exempt from contraceptive requirements. However, they must still undergo pregnancy testing as described in this section

   Exclusion Criteria:
   * Any significant acute or chronic medical illness.
   * Current or recent (within 3 months of study drug administration) gastrointestinal disease that could impact upon the absorption of study drug
   * Any other sound medical, psychiatric, and/or social reason as determined by the investigator
   * Any major surgery within 4 weeks of study drug administration.
   * Any prior GI surgery including cholecystectomy (remote history of appendectomy will not be exclusionary).
   * Current, recent (within 3 months of study drug administration), or remote history of pancreatitis.
   * Donation of blood or plasma to a blood bank or in a clinical study (except at screening visit) within 4 weeks before study drug administration.
   * Blood transfusion within 4 weeks of study drug administration. h) Inability to tolerate oral medication.
   * Inability to be venipunctured performed and/or tolerate venous access.
   * Use of tobacco- or nicotine-containing products (including, but not limited to, cigarettes, pipes, e-cigarettes, cigars, chewing tobacco, nicotine patches, nicotine lozenges, or nicotine gum) within 6 months before check-in.
   * Drug or alcohol abuse (within 2 years of study drug administration) as defined in the Diagnostic and Statistical Manual of Mental Disorders - 4th Edition, Diagnostic Criteria for Drug and Alcohol Abuse History of glucose intolerance or diabetes mellitus.
   * For females, history of chronic or recurrent urinary tract infection (UTI) (defined as 3 occurrences per year) or UTI in the past 3 months. For males, any UTI within the previous 5 years that has not been thoroughly evaluated and for which an explanation is not clear.
   * History of recurrent (defined as 3 occurrences per year) or recent vulvovaginal mycotic infections.
   * Any other sound medical, psychiatric, and/or social reason as determined by the investigator.

   Physical and Laboratory Test Findings
   1. Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECGs, or clinical laboratory determinations beyond what is consistent with the target population.
   2. Abnormal urinalysis at screening (may repeat once). If the urinalysis is abnormal on Day -1 of Period 1, continuation in the study is up to the investigator's discretion. The CRO medical monitor should be consulted.
   3. Glucosuria or hematoria at screening or Day -1 of Period 1, repeat is not permitted. d) A positive nicotine test (ie, cotinine).

   e) Abnormal liver function tests (alanine or aspartate aminotransferase [ALT or AST, respectively], or total bilirubin).

   f) Any of the following on 12-lead ECG prior to study drug administration, confirmed by repeat.

   i) PR ≥ 210 ms ii) QRS ≥ 120 ms iii) QT ≥ 500 ms iv) QTcF ≥ 450 ms g) Positive urine screen for drugs of abuse. h) Positive urine alcohol test. i) Positive blood screen for hepatitis C virus (HCV) antibody, hepatitis B surface antigen (HBsAg), or human immunodeficiency virus (HIV)-1 or HIV-2 antibodies at screening.
4. Allergies and Adverse Drug Reaction

   1. History of allergy or adverse reactions to DPP4 or SGLT inhibitors or related compounds.
   2. History of any significant drug allergy (such as anaphylaxis or hepatotoxicity).
5. Other Exclusion Criteria

   1. Prisoners or subjects who are involuntarily incarcerated.
   2. Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness.
   3. Inability to comply with restrictions and prohibited activities/treatments

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2014-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Gartner, MD, Principal Investigator — Celerion

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Open-label, randomized, single-dose, 2-treatment, 2-period crossover study in 36 healthy subjects. A single dose was administered on Day 1 and Day 8 under fasted conditions. Blood samples for the plasma pharmacokinetic analysis collected over a 60-hour interval after dosing in each period
Groups:
- Treatment AB: Treatment A: Single oral dose of 5-mg saxagliptin tablet coadministered with 10-mg dapagliflozin tablet under fasted conditions.
  Treatment B: Single oral dose of 5-mg saxagliptin/10-mg dapagliflozin FDC tablet under fasted conditions.
- Treatment BA: Treatment B: Single oral dose of 5-mg saxagliptin/10-mg dapagliflozin FDC tablet under fasted conditions.
  Treatment A: Single oral dose of 5-mg saxagliptin tablet coadministered with 10-mg dapagliflozin tablet under fasted conditions.
Period: Overall Study
Arm/Group | Treatment AB | Treatment BA
Started | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment AB | Treatment BA | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 33.6 (11.63) [19 to 53] | 32.9 (11.34) [19 to 52] | 33.3 (11.32) [19 to 53]
Age, Customized [Number; unit: Participants]
  < 65 | 18 | 18 | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 18
  Male | 10 | 8 | 18
Race/Ethnicity, Customized [Number; unit: Participants]
  BLACK/AFRICAN AMERICAN | 2 | 1 | 3
  WHITE | 16 | 17 | 33

OUTCOME MEASURES:

1. Primary Outcome: Saxagliptin Maximum Observed Concentrations (Cmax)
Description: 5-mg saxagliptin/10-mg dapagliflozin as a Fixed-dose Combination (FDC) and as Individual Tablets together in the fasted state
Time Frame: Day 1-3 (Period 1) and Day 8-10 (Period 2)
Population: Evaluable PK Population
Measure: Geometric Mean (90% Confidence Interval); unit: ng/mL
Groups:
- Treatment A: Single oral dose of 5-mg saxagliptin tablet coadministered with 10-mg dapagliflozin tablet under fasted conditions.
- Treatment B: Single oral dose of 5-mg saxagliptin/10-mg dapagliflozin FDC tablet under fasted conditions.
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 36 | 36
ng/mL | 26.2 (5.723) [24.6 to 27.8] | 25.5 (5.763) [24.0 to 27.1]
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Non-Inferiority or Equivalence — The specified bioequivalence limits (0.80, 1.25) for PK measures; p = 0.4950, ANOVA; Geometric mean ratio = 0.975, 90% CI 2-sided [0.915 to 1.038]

2. Primary Outcome: Dapagliflozin Maximum Observed Concentrations (Cmax)
Description: as for outcome 1
Time Frame: Day 1 to 3 (Period 1) and Day 8 to 10 (Period 2)
Population: Evaluable PK Population
Measure: Geometric Mean (90% Confidence Interval); unit: ng/mL
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 36 | 36
ng/mL | 142 (28.93) [132 to 153] | 141 (37.10) [132 to 152]
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Non-Inferiority or Equivalence — The specified bioequivalence limits (0.80, 1.25) for PK measures; p = 0.8650, ANOVA; Geometric mean ratio = 0.993, 90% CI 2-sided [0.932 to 1.060]

3. Primary Outcome: Saxagliptin AUC From Time 0 to Time of the Last Quantifiable Concentration (AUC[0-T])
Description: as for outcome 1
Time Frame: Day 1-3 (Period 1) and Day 8-10 (Period 2)
Population: Evaluable PK Population
Measure: Geometric Mean (90% Confidence Interval); unit: ng.h/mL
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 36 | 36
ng.h/mL | 95.9 (5.723) [90.0 to 102] | 98.0 (5.763) [92.0 to 104]
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Non-Inferiority or Equivalence — The specified bioequivalence limits (0.80, 1.25) for PK measures; p = 0.2344, ANOVA; Geometric mean ratio = 1.022, 90% CI 2-sided [0.991 to 1.054]

4. Primary Outcome: Dapagliflozin AUC From Time 0 to Time of the Last Quantifiable Concentration (AUC[0-T])
Description: as for outcome 1
Time Frame: Day 1-3 (Period 1) and Day 8-10 (Period 2)
Population: Evaluable PK Population
Measure: Geometric Mean (90% Confidence Interval); unit: ng.h/mL
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 36 | 36
ng.h/mL | 537 (5.723) [504 to 573] | 546 (5.763) [512 to 582]
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Non-Inferiority or Equivalence — The specified bioequivalence limits (0.80, 1.25) for PK measures; p = 0.2458, ANOVA; Geometric mean ratio = 1.016, 90% CI 2-sided [0.993 to 1.038]

5. Primary Outcome: Saxagliptin AUC From Time 0 Extrapolated to Infinite Time (AUC[0-inf])
Description: as for outcome 1
Time Frame: Day 1-3 (Period 1) and Day 8-10 (Period 2)
Population: Evaluable PK Population
Measure: Geometric Mean (90% Confidence Interval); unit: ng.h/mL
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 36 | 36
ng.h/mL | 97.0 (5.723) [91.1 to 103] | 99.4 (5.763) [93.3 to 106]
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Non-Inferiority or Equivalence — The specified bioequivalence limits (0.80, 1.25) for PK measures; p = 0.1947, ANOVA; Geometric mean ratio = 1.024, 90% CI 2-sided [0.993 to 1.056]

6. Primary Outcome: Dapagliflozin AUC From Time 0 Extrapolated to Infinite Time (AUC[0-inf])
Description: as for outcome 1
Time Frame: Day 1-3 (Period 1) and Day 8-10 (Period 2)
Population: Evaluable PK Population
Measure: Geometric Mean (90% Confidence Interval); unit: ng.h/mL
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 36 | 36
ng.h/mL | 553 (5.723) [518 to 591] | 561 (5.763) [525 to 599]
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Non-Inferiority or Equivalence — The specified bioequivalence limits (0.80, 1.25) for PK measures; p = 0.3191, ANOVA; Geometric mean ratio = 1.013, 90% CI 2-sided [0.992 to 1.034]

ADVERSE EVENTS:
Arm/Group | Treatment A | Treatment B
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 0/36 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No